CLINICAL TRIAL: NCT01488188
Title: A Controlled Study to Determine the Immunogenicity and Safety of Cold-adaptive Live Attenuated Influenza Vaccine (Flumist) Administered by the Nasal and Sublingual Route in Healthy Adult Volunteers
Brief Title: Immunogenicity and Safety of Live Attenuated Influenza Vaccine (Flumist) Administered by Nasal and Sublingual Route
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FM-01 V1
Record Dates: First submitted 2011-12-04; First posted 2011-12-08 (Estimated); Results first posted 2013-12-23 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-11

CONDITIONS: Healthy
Keywords: Influenza vaccine; nasal route; sublingual route; immunogenicity; safety
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Influenza vaccine-Nasal (Active Comparator): Nasal administration
  Interventions: Biological: Influenza vaccine
- Influenza vaccine -Sublingual (Active Comparator): Sublingual administration
  Interventions: Biological: Influenza vaccine

INTERVENTIONS:
Biological: Influenza vaccine — Administration of 1 dose (0.2 ml) by nasal route
  Other Names: Flumist (2011-2012)
  Arms: Influenza vaccine-Nasal
Biological: Influenza vaccine — Administration of 1 dose (0.2 ml) by sublingual route
  Other Names: Flumist (2011-2012)
  Arms: Influenza vaccine -Sublingual

SUMMARY:
Background: It is well established that live attenuated organisms can be highly effective vaccines, immune responses elicited can often be of greater magnitude and of longer duration than those produced by non-living antigens and are often able to confer protection after a single dose. Unlike killed influenza vaccine preparations injected by the parenteral route, live influenza vaccines are able to induce potent secretory (mainly IgA) antibody responses in the airway mucosae and can also evoke cell mediated responses. T cell proliferation, cytokine production, cytotoxic T cell responses and antibody-dependent cell cytotoxicity have all been elicited by live attenuated vaccines.

There has been a history of the use of live attenuated flu vaccines as safe and effective vaccines for the prevention of flu in animals and humans. Live-attenuated cold-adapted influenza vaccines have been proved to be highly efficacious to protect against clinical fly symptoms. Among these, FluMist, a nasal vaccine formulation developed by Medimmune Inc, has been approved by the US FDA. Recent side by side clinical trials have demonstrated that this nasal vaccine was significantly superior to conventional killed flu vaccine in protecting against flu symptoms.

Sublingual administration of live influenza virus at a dose lethal by the nasal route was well tolerated and did not redirect virus to the olfactory bulb. In addition, in a recent Phase I clinical study (NCT00820144) conducted in France, the sublingual administration of recombinant cholera toxin B subunit (rCTB,up to 1 mg) in healthy adult volunteers was found to be safe.

A major issue has arisen regarding the ease with which vaccines could be administered to young children, especially infants, and to elderly subjects in whom nasal vaccination has not been possible and/or approved due to difficulties of administering nasal vaccines in infants and to undesired side effects related to frequent rhinitis and sneezing episodes in elderly subjects. This study is designed to investigate the safety, tolerability and immunogenicity of a new route of administration of vaccines, using the nasal FluMist formulation as prototype vaccine.

Objectives: To evaluate the immunogenicity and safety of a nasal and sublingual influenza virus vaccine (FluMist) in healthy adult volunteers

Study design: This will be a randomized study on a total 40 subjects; each 20 subjects will receive vaccine via nasal and sublingual route, respectively

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers who are able and willing to give informed consent, following a detailed explanation of participation in the study.
* Volunteers who will be available for the duration of the study and available for scheduled and potential additional visits

Exclusion Criteria:

* Subjects with any clinically significant medical or psychiatric condition or clinically significant abnormal serum biochemistry or haematology results that, in opinion of the Investigator, preclude participation in the study.
* Female subjects who are pregnant (using urine test) or breast-feeding, or of childbearing potential and unwilling to use a reliable method of contraception (e.g. oral contraceptives or contraceptive during sexual activities such as a condom, contraceptive diaphragm, intrauterine device, hormonal contraceptive, or intercourse with a male partner who has had a vasectomy etc.) throughout the study period.
* Subjects who have known airway hypersensitivity to one of Flu vaccine excipients within 14 days prior to administration of study medication.
* Subjects who have known buccal hypersensitivity to any component of the vaccine or buffer solution used in this study, including subjects with phenylketonuria.
* Subjects with direct contact with at risk groups (e.g. patients in special care units, immuno-compromised individuals, pregnant women, children under 2 years of age and individuals over 70 years).
* Subjects with a known impairment of immune function including seropositive for HIV or those receiving (or have received in the 6 months prior to study entry) cytotoxic drugs immunosuppressive therapy (including systemic corticosteroids).
* Subjects with a significant acute febrile illness (fever of 38.0 Celsius degree or more) at time of dosing.
* Subjects who have chronic diseases: Chronic diseases will include all autoimmune and immuno-compromising conditions and any other chronic condition, which at the judgement of the Investigator, may put the subject at higher risk of side effects from the study vaccine. Conditions in the latter category might include unexplained anaemia, hepato-biliary disease, uncontrolled hypertension, subjects with prosthetic joints or heart valves, etc.
* Subjects with a current problem, based on history, with substance abuse or with a history of substance abuse
* Subjects who are currently involved in a clinical trial, have taken an investigational drug or have received investigational or licensed vaccines in the preceding 4 weeks or anticipate receiving a vaccine other than study medication during the first 4 weeks of the study
* Subjects who have known hypersensitivity to eggs or egg proteins
* Subjects who have chronic respiratory infections or syndromes
* Unable to receive oral (sublingual) administration.
* Receiving anti-viral agents.
* Subjected to contraindications and/or precautions described in drug information

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, M.D., Principal Investigator — Seoul National University Hospital; Cecil Czerkinsky, Ph.D., Principal Investigator — International Vaccine Institute
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruit volunteers at Clinical Trial Center in Seoul National University Hospital
Pre-assignment Details: Randomly group assignment
Groups:
- Influenza Vaccine -Sublingual: Sublingual administration
  Influenza vaccine : Administration of 1 dose (0.2 ml) by sublingual route
- Influenza Vaccine-Nasal: Nasal administration
  Influenza vaccine : Administration of 1 dose (0.2 ml) by nasal route
Period: Overall Study
Arm/Group | Influenza Vaccine -Sublingual | Influenza Vaccine-Nasal
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influenza Vaccine -Sublingual | Influenza Vaccine-Nasal | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25.5 (5.8) | 25.9 (4.5) | 25.7 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 13 | 8 | 21
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Passive Haemagglutination Inhibition Titer.
Description: Passive haemagglutination inhibition titer of serum at 21 days after vaccination.
Time Frame: 21 days after vaccination
Measure: Median (Full Range); unit: Titer
Arm/Group | Influenza Vaccine -Sublingual | Influenza Vaccine-Nasal
Number analyzed (Participants) | 20 | 20
Titer | 380 [5 to 560] | 440 [10 to 1120]

2. Secondary Outcome: Blood Immunoglobulin G (IgG) and Immunoglobulin A (IgA)-Antibody Secreting Cell Number to Flu Virus
Description: Flu virus-specific IgG- and IgA -antibody secreting cells per ml of blood at 7 days after vaccination
Time Frame: 7 days after vaccination
Measure: Median (Full Range); unit: cells/ml
Arm/Group | Influenza Vaccine -Sublingual | Influenza Vaccine-Nasal
Number analyzed (Participants) | 20 | 20
cells/ml | 8.85 [0.0 to 120.0] | 15.0 [0.0 to 53.8]

3. Secondary Outcome: Salivary IgA
Description: Salivary Flu-specific IgA titer at Days 21 after vaccination
Time Frame: 21 days after vaccination
Measure: Median (Full Range); unit: Titer
Arm/Group | Influenza Vaccine -Sublingual | Influenza Vaccine-Nasal
Number analyzed (Participants) | 20 | 19
Titer | 3550 [1040 to 28800] | 3600 [480 to 27200]

4. Secondary Outcome: Cell Mediated Immune Responses
Description: Interferon gamma production in peripheral blood monocyte (PBMC) after in vitro re-stimulation with influenza virus antigen at 21 days after vaccination.
Time Frame: 21 days after vaccination
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Influenza Vaccine -Sublingual | Influenza Vaccine-Nasal
Number analyzed (Participants) | 20 | 20
pg/ml | 1666 [92 to 38599] | 1743 [4 to 11674]

ADVERSE EVENTS:
Arm/Group | Influenza Vaccine -Sublingual | Influenza Vaccine-Nasal
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 3/20 | 5/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Influenza Vaccine -Sublingual (N=20) | Influenza Vaccine-Nasal (N=20)
Rhinorrhoea (General disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Mild fever (General disorders) | 2 (2) | 0 (0)
Cough (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 3 (3)
Pruitis (General disorders) | 0 (0) | 1 (1)
Constipation (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No